CLINICAL TRIAL: NCT00371306
Title: A Comparison of Glucovance (Glyburide and Metformin) to Insulin Therapy for the Treatment of Gestational Diabetes and Adult Onset Diabetes in Pregnancy
Brief Title: Comparison of Glucovance to Insulin for Diabetes During Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regional Obstetrical Consultants (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 02-078
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Gestational Diabetes; Type 2 Diabetes; Pregnancy
Keywords: Diabetes; Pregnancy
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Glyburide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Insulin versus glucovance (glyburide/metformin)

SUMMARY:
Pregnant women with gestational or Type 2 diabetes who require medication are placed in one of two groups: Insulin injections or Glucovance (oral administration). Blood glucose is checked 5 times per day, and medication adjusted by perinatologist according to glucose levels. The hypothesis is that patients will have similar or improved blood glucose control on an oral agent as compared to control on insulin.

DETAILED DESCRIPTION:
According to ACOG guidelines, patients between 24 and 28 weeks gestation will be screened with a 1 hour glucose tolerance test (GTT) by their obstetrician. Those with elevated glucose levels will undergo a 3 hour GTT. According to routine OB standards, if the blood glucose is elevated on 2 or more of 4 parameters during this test (> 95 fasting, > 180 at 1 hour, > 155 at 2 hours, >140 at 3 hours), the patient will begin receiving dietary therapy using ADA guidelines. If blood glucose levels remain 20% above a fasting of 90 & post parandial of 120 with diet alone during a period of 1-3 weeks after diagnosis, the patient will be invited to participate in this study. Type 2 diabetics who have been diagnosed prior to pregnancy will also be included. These patients may enroll in the study prior to 24 weeks gestation, entering at the time of referral. Patients who give consent for participation will be randomly assigned to either insulin therapy (the usual standard of care), or to oral Glucovance therapy (the experimental group). Glucovance will be started at 1.25mg/250mg BID. NPH & regular Insulin will be started on a 1unit/kg basis BID. Both groups will receive care according to the current standard for gestational diabetics and pregnant Type 2 diabetics. The perinatologist and diabetes educator will evaluate the blood glucose record and assess the patient's adherence to the ADA diet weekly and will determine when the insulin or Glucovance needs to be increased. If the patients in the Glucovance group continue to be poorly controlled with 4 tablets/day (5mg/500mg), the therapy will be continued and insulin will be added to the management. Statistical analysis will compare the two groups for myriad factors including vaginal versus operative deliveries, hemoglobin A1C, fructosamine, and glucose at delivery, infant birth weight, infant complications, initial infant blood glucose.

ELIGIBILITY:
Inclusion Criteria:Gestational diabetes by ACOG definition or Type 2 diabetes in pregnancy Hyperglycemia despite following ADA diet English or Spanish speaking -

Exclusion Criteria:Already requiring Insulin Serum creatinine > 1.3 or creatinine clearance < 75ml/minute Liver disease

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200
Dates: Start 2002-09; Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Maternal hemoglobin A1C at delivery
Maternal fructosamine at delivery
Maternal glucose at delivery

SECONDARY OUTCOMES:
Mode of delivery
Infant birth weight
Infant initial glucose
Infant complications

CONTACTS AND LOCATIONS:
Overall Officials: Joseph H Kipikasa, MD, Principal Investigator — Regional Obstetrical Consultants; UT Chattanooga OB-GYN Department
Locations (1):
- Regional Obstetrical Consultants, Chattanooga, Tennessee, United States